CLINICAL TRIAL: NCT01908803
Title: Proof of Concept of Single Application of AL-60371/AL-817 Otic Suspension in Treatment of Acute Otitis Media With Tympanostomy Tubes Compared to CIPRODEX® (BID for 7 Days)
Brief Title: Proof-of-Concept Study of a Single Application of an Investigational Otic Suspension in Treatment of Acute Otitis Media With Tympanostomy Tubes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Management decision
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C-13-026
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Results first posted 2015-09-24 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Acute Otitis Media
Keywords: AOMT; tympanostomy tubes; Otorrhea; anti-infective
MeSH Terms: conditions — Otitis Media | interventions — Ciprofloxacin; Dexamethasone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AL-60371/AL-817 (Experimental): AL-60371/AL-817 otic suspension, 200 μL in affected ear(s) through tympanostomy tube on Day 1 (Visit 1)
  Interventions: Drug: AL-60371/AL-817 otic suspension
- CIPRODEX (Active Comparator): Ciprofloxacin 0.3%/dexamethasone 0.1% otic suspension, 4 drops in affected ear(s) twice daily through tympanostomy tube for 7 days
  Interventions: Drug: Ciprofloxacin 0.3%/dexamethasone 0.1% otic suspension

INTERVENTIONS:
Drug: AL-60371/AL-817 otic suspension
  Arms: AL-60371/AL-817
Drug: Ciprofloxacin 0.3%/dexamethasone 0.1% otic suspension — CIPRODEX®
  Arms: CIPRODEX

SUMMARY:
The purpose of this study is to evaluate a single application of AL-60371/AL-817 Otic Suspension relative to ototopical CIPRODEX for sustained clinical cure, microbiological success, and time to cessation of otorrhea.

DETAILED DESCRIPTION:
The results at the time of the interim analysis met the futility criteria and the study was subsequently stopped.

ELIGIBILITY:
Inclusion Criteria:

* Parent or guardian: Read and sign the informed consent. When required by the Institutional Review Board, child must agree to sign an approved assent form;
* Presence of otorrhea (visible by parent or guardian) of 21 days or less in duration;
* Presence of patent tympanostomy tubes;
* Refrain from water immersion of the ears following surgery without the use of adequate ear protection during swimming, bathing, showering and other water-related activities;
* Parent or guardian: Agree to comply with the requirements of the study, administer the study medication as directed, complete required study visits, and comply with the protocol;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* NOT otorrhea-free for at least seven days following tympanostomy tube surgery;
* Menarcheal females;
* Previous otologic surgery, except tympanic membrane, within one year of study entry;
* History of/or current acute or chronic non-tube otorrhea (through existing perforation of the eardrum);
* Current acute otitis externa, malignant otitis externa, or other conditions which could interfere with evaluation of the study drug;
* Diabetic (controlled or uncontrolled);
* Use of prohibited medications;
* Other protocol-defined exclusion criteria may apply.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2013-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Manager, GCRA, Pharma, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 12 study centers located in the US.
Pre-assignment Details: Of the 84 enrolled, 14 subjects were exited as screen failures prior to randomization. This reporting group includes all randomized subjects (70).
Groups:
- AL-60371/AL-817: 200 μL in affected ear(s) through tympanostomy tube on Day 1 (Visit 1)
- CIPRODEX: Four drops in affected ear(s) twice daily through tympanostomy tube for 7 days
Period: Overall Study
Arm/Group | AL-60371/AL-817 | CIPRODEX
Started | 46 | 24
Treated | 44 (Two randomized subjects discontinued prior to receiving investigational product.) | 24
Completed | 42 | 23
Not Completed | 4 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Randomization Error | 1 | 0
Not completed — Adverse Event (pre-treatment) | 1 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized and treated subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | AL-60371/AL-817 | CIPRODEX | Total
Number analyzed (Participants) | 44 | 24 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 2.9 (2.60) | 2.4 (1.54) | 2.7 (2.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 9 | 30
  Male | 23 | 15 | 38

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Sustained Clinical Cure at Day 3 Visit
Description: A sustained clinical cure at Day 3 was attained if otorrhea was absent at the Day 3 visit and continued to be absent through the last study visit (Day 8 or Early Exit). Proportion of subjects is reported as a percentage.
Time Frame: Day 3 post-treatment up to Day 8 or Early Exit
Population: This analysis population includes all randomized subjects who received at least 1 dose of investigational product and were culture positive at the Day 1 visit in the study ear.
Measure: Number; unit: percentage of subjects
Arm/Group | AL-60371/AL-817 | CIPRODEX
Number analyzed (Participants) | 39 | 22
percentage of subjects | 38.5 | 31.8

2. Secondary Outcome: Proportion of Subjects With Microbiological Success at the Day 8 Visit
Description: Microbiological success was attained if all pre-therapy bacteria were absent in the Day 8 specimen. In a subject with no otorrhea at Day 8, eradication of pre-therapy bacteria was presumed and the subject was considered a microbiological success.
Time Frame: Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of subjects
Arm/Group | AL-60371/AL-817 | CIPRODEX
Number analyzed (Participants) | 39 | 22
percentage of subjects | NA (NA) — This outcome measure was not analyzed as a consequence of the study's early termination. | NA (NA) — This outcome measure was not analyzed as a consequence of the study's early termination.

3. Secondary Outcome: Median Time (in Days) to Cessation of Otorrhea
Description: Median time (in days) to the cessation of otorrhea (ie, otorrhea was absent) was calculated as the number of days from the Day 1 (Visit 1) to the absence of otorrhea in the affected ear(s) as recorded by the parent/guardian via the twice-daily diary. Cessation of otorrhea was defined as ending on the first day that otorrhea was absent from the affected ear(s) and remained absent for any/all subsequent diary entries.
Time Frame: Time to event, up to Day 8
Population: as for outcome 1
Measure: Median (Standard Error); unit: days
Arm/Group | AL-60371/AL-817 | CIPRODEX
Number analyzed (Participants) | 39 | 22
days | NA (NA) — This outcome measure was not analyzed as a consequence of the study's early termination. | NA (NA) — This outcome measure was not analyzed as a consequence of the study's early termination.

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected for the duration of subject participation in the study (8-10 days). AEs are reported as pre-treatment and treatment-emergent.
Description: An AE was defined as any untoward medical occurrence in a subject who is administered a study treatment regardless of whether or not the event has a causal relationship with the treatment. AEs were obtained as solicited comments from the study patients and as observations by the Investigator as outlined in the study protocol.
Groups:
- Pre-treatment: Includes all subjects prior to administration of study medication
- AL-60371/AL-817: Includes all subjects administered a dose of AL-60371/AL-817
- CIPRODEX: Includes all subjects administered a dose of CIPRODEX®
Arm/Group | Pre-treatment | AL-60371/AL-817 | CIPRODEX
Serious Adverse Events (participants affected / at risk) | 0/84 | 0/44 | 0/24
Other Adverse Events (participants affected / at risk) | 0/84 | 3/44 | 1/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-treatment (N=84) | AL-60371/AL-817 (N=44) | CIPRODEX (N=24)
Otitis media acute (Infections and infestations) | 0 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.